CLINICAL TRIAL: NCT01244048
Title: Intervention With n3 LC-PUFA-supplemented Yogurt: Effects on Cardiovascular Risk Factors and Inflammatory Biomarkers
Brief Title: Intervention With n3 LC-PUFA-supplemented Yogurt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Proffessor Dr. G. Jahreis, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LSEP H35_08
Record Dates: First submitted 2010-11-16; First posted 2010-11-19 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Moderate Hypertriacylglycerolemic Subjects
Keywords: n3 LC-PUFA, yoghurt, inflammatory markers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: n3 long chain polyunsaturated fatty acids — Group 1 (placebo) Group 2 (0.8 g n3 LC-PUFA/d in 125 g yoghurt) Group 3 (3 g n3 LC-PUFA/d in 200 g yoghurt)

SUMMARY:
The effective dosage of a n3-LC-PUFA intervention (with n3 LC-PUFA-enriched yoghurt) on the modulation of cardiovascular risk factors and inflammatory biomarkers were determined.

DETAILED DESCRIPTION:
Fifty three mildly hypertriacylglycerolemic subjects (TAG ≥ 150 mg/dL (1.7 mmol/L)) participated on the placebo-controlled, double-blind, parallel designed study.

The subjects consumed placebo yoghurt (1), or n3 LC-PUFA-enriched yoghurt (0.8 g n3 LC-PUFA/d (2), 3 g n3 LC-PUFA/d (3)) for 10 weeks.

Blood samples were taken at the beginning and at the end of the period.

Parameters:

* Blood lipids (total cholesterol, HDL, LDL, triacylglycerols)
* Fatty acid distribution of plasma lipids (PL) and erythrocyte membranes (EM)
* Concentrations of eicosanoids (PGs, HETEs)
* Production of ex vivo stimulated cytokines by T cells
* SNPs in the CD36 genotype

ELIGIBILITY:
Inclusion Criteria:

* hypertriacylglycerolemic subjects (TAG: ≥ 150 mg/dl (1.7 mmol/l))

Exclusion Criteria:

* patients receiving blood-diluting and lipid-lowering medications or glucocorticoids
* patients suffering from gastrointestinal or metabolic diseases (e.g., diabetes mellitus, hyper- and hypothyroidism) and hypercholesteremic patients with familial previous impacts
* patients taking dietary supplements (e.g., fish oil capsules, vitamin E) or having either known allergies or foodstuff indigestibility
* further exclusion criteria: smoking, high sportive activity or daily alcohol intake

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Blood lipids (total cholesterol, HDL, LDL, triacylglycerols) | change from baseline after 10 weeks
  change from baseline after 10 weeks
  Group 1: placebo Group 2: 0.8 g n3 LC-PUFA/125 g yoghurt per day Group 3: 3 g n3 LC-PUFA/200 g yoghurt per day

SECONDARY OUTCOMES:
fatty acid distribution in plasma lipids and erythrocyte membranes, eicosanoids in plasma, production of ex vivo stimulated cytokines by T cells, SNPs on CD36 genotype | change from baseline after 10 weeks
  change from baseline after 10 weeks
  Group 1: placebo Group 2: 0.8 g n3 LC-PUFA/125 g yoghurt per day Group 3: 3 g n3 LC-PUFA/200 g yoghurt per day

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Department of Nutrition, University Jena
Locations (1):
- University of Jena, Institute of Nutrition, Department of Nutritional Physiology, Jena, Germany

REFERENCES:
- [Derived] Dawczynski C, Massey KA, Ness C, Kiehntopf M, Stepanow S, Platzer M, Grun M, Nicolaou A, Jahreis G. Randomized placebo-controlled intervention with n-3 LC-PUFA-supplemented yoghurt: effects on circulating eicosanoids and cardiovascular risk factors. Clin Nutr. 2013 Oct;32(5):686-96. doi: 10.1016/j.clnu.2012.12.010. Epub 2012 Dec 28. PMID 23332800